CLINICAL TRIAL: NCT04772833
Title: Observational, Multicenter, Cross-sectional Study at National Level to Analyze the Histopathological, Ultrastructural and Microbiological Findings Obtained in Autopsies of Patients Who Died Due to COVID-19 in Spain
Brief Title: Spanish Study to Analyze the Histopathological, Ultrastructural and Microbiological Findings Obtained in Autopsies of Patients Who Died Due to COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: Spanish Society of Infectious Diseases and Clinical Microbiology (Unknown); Spanish Society of Pathological Anatomy (Unknown)
Responsible Party: Sponsor
Other Study IDs: NECROVID
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Covid19
Keywords: COVID-19; Autopsy; Histopathological findings; Ultrastructural findings; Microbiological findings
MeSH Terms: conditions — COVID-19 | interventions — Autopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The following samples will be collected:
  * Laboratory of Pathology:
    1. Histopathological study: the samples collected from all the organs and tissues will be fixed in 10% formaldehyde.
    2. Electron Microscopy study: lung, myocardium, kidney and muscle samples they will be fixed in Glutaraldehyde for study by Electron Microscopy.
  * Biobank: 2 samples will be collected - the first sample will be in fresh and the second one will be preserved with RNAlater.
  * Microbiology Laboratory: respiratory secretions and tissue sample will be collected for bacterial and fungal cultures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Autopsy group: Patients with COVID-19 infection confirmed by PCR, whose death is related to active COVID-19 infection or its complications.
  Interventions: Other: Autopsy

INTERVENTIONS:
Other: Autopsy — The subjects deceased will undergo an autopsy to analyze the histopathological, ultrastructural and microbiological findings, related to the COVID-19 disease.

SUMMARY:
The aim of this study is prospectively analyzing the histopathological, ultrastructural and microbiological findings from autopsies performed on patients with COVID-19.

DETAILED DESCRIPTION:
The aim of this study is to increase the knowledge of the pathogenic mechanisms of the COVID-19 disease, that will allow us to improve the design of clinical and therapeutic strategies against the disease. This is the tool to improve the prognosis of patients with COVID-19.

The performance of systematic and regulated autopsies can help to manage it. However, despite the need to generate this knowledge and the strong impact on mortality caused by the COVID-19 pandemic, the evidence from post-mortem studies is very limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COVID-19 infection confirmed by PCR.
* Death related to active infection by COVID-19 or its complications.
* Informed consent given by the subject's relatives to perform an autopsy according to the autonomous community requirements.
* Informed consent given by the subject's relatives for the inclusion of samples in the Biobank.

Exclusion Criteria:

* COVID-19 infection diagnosed exclusively by serological methods.
* Advanced or terminal chronic disease.
* Inadequate security level of the autopsy room.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with COVID-19 infection confirmed by PCR, whose death is related to active COVID-19 infection or its complications.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Histopathological and ultra-structural findings | End of autopsy
  To analyze the histopathological and ultra-structural findings obtained in complete and systematic autopsies of patients who died due to COVID-19.

SECONDARY OUTCOMES:
Molecular characterization | End of autopsy
  To analyze the presence and molecular characterization of COVID-19 in the different organs obtained in autopsies of patients deceased by COVID-19.
Hidden pulmonary superinfections | End of autopsy
  To evaluate the frequency of hidden pulmonary superinfections (bacterial and fungal disease) in patients who died due to COVID-19.
Histopathological / ultra-structural findings and clinical / biological expression correlation | End of autopsy
  To correlate the histopathological and ultra-structural findings obtained in autopsies with the clinical and biological expression of patients who died due to COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Rivero Román, MD, Principal Investigator — Spanish Society of Infectious Diseases and Clinical Microbiology. Reina Sofía University Hospital.; Teresa Hermida Romero, MD, Study Chair — Spanish Society of Pathological Anatomy. A Coruña University Hospital; Xavier Matias--Guiu Guia, MD, Study Chair — Spanish Society of Pathological Anatomy. Bellvitge University Hospital; Jordi Vila Estapé, MD, Study Chair — Spanish Society of Infectious Diseases and Clinical Microbiology. Barcelona Clinic University Hospital.
Locations (10):
- Spain (10):
  - Marqués de Valdecilla University Hospital, Santander, Cantabria
  - Puerta de Hierro University Hospital, Majadahonda, Madrid
  - Navarra University Hospital, Pamplona, Navarre
  - Barcelona Clinic University Hospital, Barcelona
  - Reina Sofía University Hospital, Córdoba
  - Ramón y Cajal University Hospital, Madrid
  - Fundación Jiménez Díaz University Hospital, Madrid
  - 12 de Octubre University Hospital, Madrid
  - Virgen del Rocío University Hospital, Seville
  - Araba University Hospital, Vitoria-Gasteiz, Álava

IPD SHARING:
Plan to Share IPD: Yes
All the information collected will be shared with other researchers under request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The information will be shared after the results are published in the concerning papers.
Access Criteria: The information will be shared upon request, contacting uicec@imibic.org.